CLINICAL TRIAL: NCT05679518
Title: Managing Fear of Cancer Progression Metacognition-based Vs Supportive-expressive Based Approaches: A Randomized Controlled Trial
Brief Title: Managing Fear of Cancer Progression Metacognition-based Vs Supportive-expressive Based Approaches
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Wendy Wing Tak Lam, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW22-036
Record Dates: First submitted 2022-12-19; First posted 2023-01-11 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Advanced or Metastatic Cancer; Fear of Cancer Progression; Metacognition-based Intervention; Supportive-expressive Based Intervention; Psychooncology
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: The investigators will use a block randomization structure with randomly permuted block sizes of 3 and 6 to ensure a close balance of the numbers in each arm. Randomization (by a statistician) occurs prior to eligible patients attending the clinic to minimize opportunities for selection bias.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, care provider, and outcomes assessor are masked in terms of not knowing to which condition the participants will be randomized until after the completion of the baseline assessment. The outcomes assessor will break the envelope for the next eligible participant indicating if that participant is to be allocated to ConquerFear or CALM or control arms.
  The participants are masked in terms of not knowing that the interventions (i.e. Conquer fear and CALM) are hypothesized to yield larger effects than the other (i.e. control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ConquerFear intervention (Experimental): Participants in the ConquerFear intervention group will receive a manualized intervention, consisting of 6 therapist-led individual sessions.
  Interventions: Behavioral: ConquerFear intervention
- CALM intervention (Experimental): Participants in the CALM intervention group will receive a semi-structured, manualized, individual psychotherapy intervention consisting of 3-6 individual therapy sessions.
  Interventions: Behavioral: CALM intervention
- Basic Cancer Care (Active Comparator): Basic Cancer Care serves as an active comparator and is not developed specifically to target fear of cancer recurrence through modifying participants' cognitive beliefs. Participants in this arm will receive 6 individual sessions including 2 relaxation training sessions, 2 dietetic consultation sessions, and 2 exercise sessions, which will be led by a trained therapist, a registered dietitian, and an exercise physiologist, respectively.
  Interventions: Behavioral: Basic Cancer Care

INTERVENTIONS:
Behavioral: ConquerFear intervention — ConquerFear is a manualized intervention, consists of six individual sessions over 10 weeks. The key goals of this intervention are the following: (1) teach strategies for controlling worry and excessive threat monitoring, (2) modify underlying unhelpful beliefs about worry, (3) develop appropriate monitoring and screening behaviours, (4) encourage acceptance of the uncertainty brought about by a cancer diagnosis, and (5) clarify values and encourage engagement in values-based goal setting (19). Each session will last 60-90 minutes and be delivered by a trained therapist. After each session, participants will be given home-based exercises to practice the skills learned in the sessions. With the uncertainty surrounding the COVID-19 pandemic, instead of face-to-face sessions only, a hybrid mode of intervention delivery will be used by offering participants the choice of face-to-face or online sessions.
  Arms: ConquerFear intervention
Behavioral: CALM intervention — CALM is a semi-structured, manualized, individual psychotherapy intervention designed for patients with advanced cancer. It includes 3-6 individual therapy sessions, with each approximately lasts 45-60 minutes, delivered over 3-6 months. The sessions cover 4 domains: 1) symptom management and communication with health care providers; 2) changes in self and relations with close others; 3) sense of meaning and purpose; and 4) the future and mortality. All modules will be addressed with each patient, but the sequencing and time devoted to each domain can be varied, based on the concerns that are most relevant to each patient.
  Arms: CALM intervention
Behavioral: Basic Cancer Care — Basic Cancer Care intervention for the control arm was developed to help cancer survivors with health maintenance in long-term through providing comprehensive lifestyle guidance. The intervention incorporates relaxation training, dietary and physical fitness consultations with the key goals to (1) teach relaxation techniques, (2) offer personalized diet and physical activity advice, and (3) enhance survivors' perceived control over illness, thereby leading to better adjustment to cancer. Similar to the ConquerFear intervention, Basic Cancer Care intervention consists of 6 individual sessions over 10 weeks. Each session will last 60-90 minutes and be delivered by a trained therapist, a registered dietitian, and an exercise physiologist, respectively. A hybrid mode of intervention delivery will be also used by offering participants the choice of face-to-face or online sessions.
  Arms: Basic Cancer Care

SUMMARY:
The present study aims to conduct a randomized controlled trial to assess the effect of CALM intervention and ConquerFear intervention on fear of cancer progression among Chinese patients diagnosed with advanced cancer.

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted to assess the effect of CALM intervention and ConquerFear intervention on fear of cancer progression among Chinese patients diagnosed with advanced cancer.

The aims are to test:

1. the direct effect of CALM intervention or ConquerFear intervention on fear of cancer progression, and
2. the indirect effect of ConquerFear intervention on fear of cancer progression through its effect on maladaptive metacognition.

Primary hypothesis:

1. Patients receiving CALM intervention or ConquerFear intervention, compared to those receiving a basic cancer care intervention will show a reduction in fear of cancer progression.
2. Both CALM intervention and ConquerFear intervention will be equally effective in reducing fear of cancer progression.
3. Given ConquerFear intervention aims to modify unhelpful metacognitive beliefs, there will be an indirect effect of ConquerFear intervention on fear of cancer progression through its effect on maladaptive metacognition.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese- or Mandarin-speaking Chinese patients recently diagnosed with advanced or metastatic (i.e. stage III or IV) cancer
* are the age of 18 years or above

Exclusion Criteria:

* Patients with major communication difficulties
* are being unwilling or unable to commit 6 psychotherapy sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Fear of Progression | Baseline, the immediate post-intervention, 3-months post-intervention and 6-months post-intervention
  The 12-item short version of the Fear of Progression Questionnaire (FoP-Q-SF) will be used to assess the change in total score of fear of caner progression. Each item of the FoP-Q-SF is rated on 5-point Likert scales anchored at 1 (Never) to 5 (very often). Higher scores indicate higher levels of fear of cancer progression. Total scores range from 12 to 60. A cutoff of 24-33 was used to suggest subthreshold level of fear of progression and a score of 34 or greater suggest high levels of fear of progression.

SECONDARY OUTCOMES:
Metacognitions | Baseline, the immediate post-intervention, 3-months post-intervention and 6-months post-intervention
  The 30-items Metacognitions questionnaire (MCQ-30) will be used to assess the change of metacognitive beliefs.Each item is rated on a 4-point Likert scale with a total score ranging from 30 to 120. High scores indicate a more maladaptive metacognitive style.
Depression | Baseline, the immediate post-intervention, 3-months post-intervention and 6-months post-intervention
  Change in total scores of depression will be assessed using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 score can range from 0 to 27, with higher scores indicative of a higher level of depression. The PHQ-9 is a reliable and valid 9-item measure of depression that has been used widely in advanced cancer patients.
Death anxiety | Baseline, the immediate post-intervention, 3-months post-intervention and 6-months post-intervention
  Change in total scores of death anxiety will be assessed by the 15-item Death and Dying Distress Scale (DDDS). The DDS score can range from 0 to 90, with higher scores indicative of a higher level of death anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Wing Tak Lam, PhD, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (4):
- Hong Kong (4):
  - Queen Mary Hospital-Department of Obstetrics & Gynaecology, Hong Kong
  - Queen Mary Hospital-Department of Oncology, Hong Kong
  - Queen Mary Hospital-Department of Surgery, Hong Kong
  - Tung Wah Hospital-Department of Surgery, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available from the PI upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Information will be available from the PI upon reasonable request. The author to review requests is the PI.